CLINICAL TRIAL: NCT03796780
Title: Comparison of Effects of Extra-virgin and Refined Olive Oil Consumption on Plasma Lipids and Inflammatory Markers in Patients Undergoing Coronary Angiography
Brief Title: Comparison of Extra-Virgin and Refined Olive Oil on Some Cardiovascular Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Javad Nasrollahzadeh (Other)
Collaborators: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Javad Nasrollahzadeh, Investigator in Clinical Nutrition, Shahid Beheshti University
Organization: Shahid Beheshti University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 425
Record Dates: First submitted 2018-12-29; First posted 2019-01-08 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Cardiovascular Risk Factor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extra-Virgin Olive Oil (Active Comparator): Daily consumption of 25 mL Extra-Virgin Olive Oil for 6 weeks
  Interventions: Dietary Supplement: Extra-Virgin Olive Oil
- Refined Olive Oil (Placebo Comparator): Daily consumption of 25 mL Refined Olive Oil for 6 weeks
  Interventions: Dietary Supplement: Refined Olive Oil

INTERVENTIONS:
Dietary Supplement: Extra-Virgin Olive Oil — Daily consumption of 25 mL Extra-Virgin Olive Oil in adjunct to medical treatment for 6 weeks
  Arms: Extra-Virgin Olive Oil
Dietary Supplement: Refined Olive Oil — Daily consumption of 25 mL Refined Olive Oil in adjunct to medical treatment for 6 weeks
  Arms: Refined Olive Oil

SUMMARY:
Consumption of extra-virgin olive oil has beneficial effects on cardiovascular risk factors. The purpose of this study is to compare the effects of extra-virgin olive oil and refined olive oil, in adjunct to conventional medical treatment, in improving liver enzymes, plasma lipid profile and inflammatory markers in patients with cardiovascular risk factors.

DETAILED DESCRIPTION:
A randomized placebo controlled clinical trial will be conducted in Rajaie Cardiovascular Center in Tehran, Iran. After review of the inclusion and exclusion criteria and explanation of the design of the study, written consent form will be completed. The participants are 40 eligible patients, aged 20-75 years. Intervention group will be received 25 mL/d extra-virgin olive oil and control group will be received 25 mL/d refined olive oil for 6 weeks. Fasting blood sample will be taken to measure lipid profile, liver enzymes and inflammatory markers (Interleukine-6 [IL-6] and Interleukine-10 [IL-10] and C-Reactive Protein [CRP]).

ELIGIBILITY:
Inclusion Criteria:

1. patients with at least one of the cardiovascular risk factors (hypertension, hyperlipidemia, diabetes mellitus) candidate for angiography
2. willing to participation in the study

Exclusion Criteria:

1. Continuous consumption of any supplement with anti-inflammatory or antioxidant properties such as Omega-3, vitamin E, vitamin C and Selenium in last month
2. َChronic kidney disease stage 5
3. Any change in disease treatment plan such as change in type and dose of lipid lowering drugs or surgical operation

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Interleukin-6 (IL-6) | 6 week
  change in plasma level of interleukin-6 (IL-6) in pg/mL from baseline at week-6

SECONDARY OUTCOMES:
plasma lipid profile | 6 week
  change in plasma level of lipoproteins in mg/dL from baseline at 6 week
plasma liver enzymes (SGOT & SGPT) | 6 week
  change in plasma level of liver enzymes (SGOT & SGPT) in mg/dL from baseline at 6 week
Interleukin-10 (IL-10) | 6 week
  Change in plasma level of interleukin-10 (IL-10) in pg/mL at baseline and week-6
C reactive protein (CRP) | 6 week
  Change in plasma level of C reactive protein (CRP) in mg/dL from baseline and week-6

CONTACTS AND LOCATIONS:
Overall Officials: Javad Nasrollahzadeh, Ph.D, Study Chair — Shahid Beheshti University of Medical Sciences
Locations (1):
- Rajaei Cardiovascular, Medical & Research Center, Tehran, Iran

REFERENCES:
- [Derived] Khandouzi N, Zahedmehr A, Nasrollahzadeh J. Effect of polyphenol-rich extra-virgin olive oil on lipid profile and inflammatory biomarkers in patients undergoing coronary angiography: a randomised, controlled, clinical trial. Int J Food Sci Nutr. 2021 Jun;72(4):548-558. doi: 10.1080/09637486.2020.1841123. Epub 2020 Oct 29. PMID 33121297